CLINICAL TRIAL: NCT03230708
Title: A Phase I/II Clinical Trial Study on Autologous Erythrocytes Derived Microparticles Packaging Methotrexate Peritoneal Perfusion in the Treatment of Malignant Ascites
Brief Title: Clinical Study of Autologous Erythrocytes Derived MPs Packaging MTX Peritoneal Perfusion to Treat Malignant Ascites
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hui ting Xu，MD (Other)
Responsible Party: Sponsor-Investigator, Hui ting Xu，MD, Deputy Chief Physician, Hubei Cancer Hospital
Organization: Hubei Cancer Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP-FS-002
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Malignant Ascites
Keywords: Microparticles; Erythrocytes; Methotrexate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erythrocytes derived MPs containing MTX (Experimental): Suspension of erythrocytes derived MPs containing MTX, qd×6, 6 units MPs a time , Two courses.
  Interventions: Other: Erythrocytes derived MPs containing MTX
- convention drugs (Active Comparator): Chemotherapeutic drugs, biologicals or traditional Chinese medicine.Dosage form, dosage, frequency and duration according to respective medicine instructions.
  Interventions: Drug: convention drugs

INTERVENTIONS:
Other: Erythrocytes derived MPs containing MTX — General conventional treatment and peritoneal drainage, additional peritoneal perfusion with erythrocytes derived MPs containing MTX
  Other Names: Systemic therapy
  Arms: Erythrocytes derived MPs containing MTX
Drug: convention drugs — according to usage method of drugs
  Other Names: Systemic therapy
  Arms: convention drugs

SUMMARY:
This study makes an observation over the objective response rate of autologous erythrocytes derived microparticles packaging methotrexate peritoneal perfusion and systemic therapy combination in the treatment of malignant ascites. All the participants will randomly receive the treatment of autologous erythrocytes derived microparticles packaging methotrexate peritoneal perfusion and systemic therapy combination or convention drugs peritoneal perfusion and systemic therapy combination.

DETAILED DESCRIPTION:
As a drug carrier, erythrocytes have their own advantages, such as high biocompatibility, high immune compatibility, simple structure and easy access. In this study, microparticles released from erythrocytes are used as the carrier of chemotherapy drugs and effectively kill tumor cells in malignant ascites. These microparticles can easily reach the tumor site and bring the drug into tumor cells, which can overcome the two main problems in normal chemotherapy: damage to normal cells and drug resistance of tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* 18 and ≤ 80 years of age
* Histological confirmed gastric cancer, colorectal cancer, or ovarian cancer, tumor cells were detected by exfoliative cytology of peritoneal effusion, refractory or recurrent ascites of ovarian cancer were required, other kinds of cancer were not limited
* Vital signs were stable, Karnofsky ≥ 70, life expectancy of more than 3 months
* The hematopoietic function of bone marrow was normal without bleeding tendency (INR < 1.5), blood routine examination: HGB ≥ 90 g/L, WBC > 4.0 × 10^9/L (NEU ≥ 1.5 × 10^9/L), PLT ≥ 80 × 10^9/L
* Liver function: STB ≤ 1.5 ULN, AST and ALT≤ 2.5 ULN (if the abnormity of liver function was mainly caused by tumor invasion, AST and ALT ≤ 5 ULN), ALP ≤ 1.5 ULN
* Renal function: BUN and Cr ≤ 1.5 ULN, CCr ≥ 50mL/min
* ECG and blood glucose level were normal
* Patients or family members agreed to participate in the study and signed informed consent
* No other serious heart and lung disease, etc.

Exclusion Criteria:

* Pregnant or lactating women
* Allergic constitution and multi-drug allergy
* Serious heart, lung, liver and kidney dysfunction, decompensated heart, lung, kidney, liver and other major organs dysfunction or failure, poor blood glucose control, chemotherapy intolerance, combined intestinal obstruction
* Concurrent severe infection
* HIV positive, HBsAg and HBV DNA copy number positive (quantitative detection ≥ 1000 cps/mL), chronic hepatitis C blood screening positive (HCV antibody positive)
* Cognitive impairment or poor chemotherapy compliance determined by investigator
* Less than 4 weeks from the last clinical trial
* Unsuitable for clinical trials determined by investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2018-02-01 (Estimated)

PRIMARY OUTCOMES:
ORR, Objective Response Rate | From assignment of the first subject to 2 months later after the last participant is recruited.
  The percentage of subjects with total number of Complete Response (CR) + total number of Partial Response (PR)

SECONDARY OUTCOMES:
DCR, Disease Control Rate | From assignment of the first subject to 2 months later after the last participant is recruited.
  DCR is defined as the percentage of subjects whose best response was not Progressive Disease (PD) according to Response Evaluation Criteria in Solid Tumors (RECIST) (= total number of Complete Response (CR) + total number of Partial Response (PR) + total number of Stable Disease (SD)

CONTACTS AND LOCATIONS:
Overall Officials: Yan li Nie, MD, Principal Investigator — Hu bei CH
Locations (1):
- Hui ting Xu, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No